CLINICAL TRIAL: NCT07330830
Title: Study of PNPLA3 Genetic Polymorphisms in Patients With Non-Alcoholic Fatty Liver Disease in an Ultramarine Population
Brief Title: Study of PNPLA3 Genetic Polymorphisms in Patients With Non-Alcoholic Fatty Liver Disease in an Ultramarine Population (AdipoDROMExpo)
Acronym: AdipoDROMExpo
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH2_2025/04
Record Dates: First submitted 2025-11-14; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: MASLD/MASH (Metabolic Dysfunction-Associated Steatotic Liver Disease / Metabolic Dysfunction-Associated Steatohepatitis)
Keywords: MASLD; MASH; PNPLA3; genetic polymorphism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA library for search of genetic polymorphism collected in 2 EDTA tubes of 8 mL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic Dysfunction Associated Liver Disease (MASLD) is associated with metabolic syndrome, and PNPLA3 variants are known to be implicated in intrahepatic lipid accumulation and linked to lipotoxicity. Analysis of PNPLA3 polymorphisms in an overseas territories population of MASLD would be interesting to describe their profile susceptibility to develop Metabolic dysfunction associated steatohepatitis (MASH).

DETAILED DESCRIPTION:
Metabolic dysfunction associated liver disease (MASLD) is a significant public health concern worldwide with a complex etiology attributed to behavioural, environmental, and genetic causes. The worldwide prevalence of MASLD is estimated to be 32.4% and constantly rising.

Several studies suggest differences in the prevalence and severity of MASLD by race or ethnicity, which may be linked to differences in lifestyle, diet, metabolic comorbidity profile, and genetic background, among others.

Race/ethnicity research is essential as it can provide valuable information regarding biological and genetic differences among people with similar cultural, dietary, and geographical backgrounds.

There is ample epidemiological evidence on the role of genetic susceptibility in MASLD, mainly from studies showing the clustering of MASLD cases among families and observing differences in the prevalence and severity of MASLD among ethnicities.

The Overseas territories population is predominantly of African descent due to slave trade of population from sub-Saharan Africa between the seventeenth and nineteenth centuries. They have also been a mixture from Europeans and Indians. Indian are descents from Latin America, initially present on the territories, and from Asia, after the abolition of slavery. Data about MASLD in Overseas territories are scarce. To our knowledge, one study reported the prevalence of MASLD in Caribbean and Hispanic populations resident in the United States compared with Hispanic residents in Latin America (Kallwitz 2015). In the later study, rates of MASLD were significantly lower in persons with Caribbean origin than those of Latin America heritage.

Genetic susceptibility variations may partially explain the heterogeneity observed in the MASLD prevalence/incidence estimates from different geographical regions and the variability in disease severity among individuals. Genetic factors have been suggested as one of the underlying causes of racial/ethnic differences in susceptibility to MASLD.

Among the building blocks of metabolic syndrome, type 2 diabetes and obesity have been significantly associated with an increased risk of MASH with more severe progression to cirrhosis or liver cancer.

However, in overseas, the prevalence of type 2 diabetes (10%), high blood pressure (28%), or obesity (30%) are among the highest in France.

PNPLA3 expression is implicated in intrahepatic lipid accumulation and is associated with lipotoxicity and the more severe phenotypes, including fibrosis and carcinogenesis. Therefore, in this study, PNPLA3 polymorphisms will be analysed to evaluate the profile of MASLD patients in overseas territories. A biological sample will be taken to analyse PNPLA3 polymorphisms in DROMSteatExpo study.

ELIGIBILITY:
IInclusion Criteria

-Adult patients (≥18 years old) seen in consultation or hospitalized in the Hepato-Gastroenterology Departments of the University Hospitals of Guadeloupe, French Guiana, and Réunion Island, with a diagnosis of MASLD.

MASLD is defined as evidence of hepatic steatosis associated with overweight/obesity, type 2 diabetes, or metabolic syndrome according to ATP III (2005) criteria.

* Patients affiliated with, or beneficiaries of, a social security scheme.
* Free, informed, and written consent obtained from the participant and signed by both the participant and the investigator (no later than the day of inclusion and prior to any procedure required by the study).

Exclusion Criteria:

* Patients under 18 years of age.
* Patients unable to provide informed consent; so-called vulnerable populations (individuals under guardianship, judicial protection, etc.).
* Presence of another cause of chronic liver disease, including:

Viral hepatitis (B, C, or E)

Primary biliary cholangitis or primary sclerosing cholangitis

Autoimmune hepatitis

Wilson's disease

Hemochromatosis

Alpha-1 antitrypsin deficiency

Alcoholic liver disease, or daily alcohol consumption >30 g/day for men or >20 g/day for women

-Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective longitudinal multicentric study
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2027-11-26 (Estimated); Study Completion 2027-11-28 (Estimated)

PRIMARY OUTCOMES:
Allele frequencies of PNPLA3 variants | Baseline (inclusion visit).
  The primary outcome is the allele frequencies of PNPLA3 gene variants in patients with Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) from the overseas population. Genotyping will be performed on DNA extracted from patient blood samples, and the frequency of each allele will be reported as the proportion of participants carrying the variant.

SECONDARY OUTCOMES:
Distribution of MASLD Clinical Stages at Baseline | Baseline (inclusion visit).
  The distribution of Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) clinical stages at baseline will be assessed by physician clinical evaluation. Participants will be classified into clinical categories including simple steatosis and non-alcoholic steatohepatitis (NASH). The outcome will be reported as the number and percentage of participants in each clinical stage.
Distribution of Liver Fibrosis Stages Assessed by Imaging at Baseline | Baseline (inclusion visit).
  Liver fibrosis stage will be assessed at baseline using imaging-based liver stiffness measurements (e.g., transient elastography, magnetic resonance elastography, or MRI-based techniques, as available at participating centers). Fibrosis stages will be categorized according to standard fibrosis stages (F0-F4). The outcome will be reported as the number and percentage of participants in each fibrosis stage.
Distribution of MASLD Severity Based on Laboratory Biomarkers at Baseline | Baseline (inclusion visit).
  MASLD severity will be assessed at baseline using laboratory biomarkers, including liver enzymes (e.g., ALT, AST) and metabolic parameters. Results will be categorized according to predefined clinical thresholds. The outcome will be reported as the number and percentage of participants within each severity category.

CONTACTS AND LOCATIONS:
Overall Officials: Moana Gelu-Simeon, MD PhD, Study Chair — CHU de la Guadeloupe
Locations (3):
- Centre Hospitalier Universitaire de la Guyane, Cayenne, French Guiana
- CHU de la Guadeloupe, Pointe-à-Pitre, Guadeloupe
- Centre Hospitalier Universitaire de la Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: Undecided